CLINICAL TRIAL: NCT06737653
Title: Effect of Antimicrobial Gel With Postbiotics, Lactoferrin, Aloe Barbadensis Leaf Juice Powder and Sodium Hyaluronate on Palatal Mucosa Wound Healing: a Randomized Clinical Trial
Brief Title: Palatal Mucosa Wound Healing Following Antimicrobial Gel Application
Acronym: BIOR_01
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea Pilloni MD DDS MS, Principal Investigator, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0151/2023
Record Dates: First submitted 2024-12-11; First posted 2024-12-17 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2024-12

CONDITIONS: Wound Healing; Palate; Wound; Hyaluronic Acid
Keywords: wound healing; palatal mucosa; hyaluronic acid; lactoferrin; postbiotics; aloe
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Split-mouth design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- antimicrobial gel containing postbiotics, lactoferrin, aloe barbadensis leaf juice powder and sodium (Experimental): antimicrobial gel containing postbiotics, lactoferrin, aloe barbadensis leaf juice powder and sodium hyaluronate
  Interventions: Device: Gel containing postbiotics, lactoferrin, aloe barbadensis leaf juice powder and sodium hyaluronate
- Placebo group (Placebo Comparator): Placebo gel
  Interventions: Device: Placebo gel

INTERVENTIONS:
Device: Gel containing postbiotics, lactoferrin, aloe barbadensis leaf juice powder and sodium hyaluronate — The gel will be applied until the wound is filled with the gel, which will be left undisturbed for 5 min.
  Arms: antimicrobial gel containing postbiotics, lactoferrin, aloe barbadensis leaf juice powder and sodium
Device: Placebo gel — The gel will be applied until the wound is filled with the gel, which will be left undisturbed for 5 min.
  Arms: Placebo group

SUMMARY:
The present study will be a prospective, randomized, triple-blind, split-mouth, clinical trial.

The study timeline will be include seven total visits. After a screening/study enrolment visit, a wounding surgery visit (Day 0) will be schedule. On Day 0, one standardized wound will be created on each side of the palate (DFGG required for root coverage procedure). Each side of the palate randomly received either antimicrobial gel (treatment group) or placebo (control group) at day 0, 1 and 3.

The patients, an experienced periodontist who performed the surgical procedures and the clinical examiners will be blinded to treatment allocation.

Clinical healing response and patient related outcome measures (PROMs) will be evaluated on postoperative Day 1, 3, 7, 14, 21 and 30.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 38 years (age limits based on evidence of delayed wound healing in older adults, Engeland et al., 2006);
* full-mouth plaque score and full-mouth bleeding score ≤ 15% at study entry;
* adequate anteroposterior arch length for required wound size and spacing;
* able to easily tolerate maxillary impression making and use of palatal template;
* patients required at least two root coverages procedures in one tooth in different sextants with DFGG;
* palate with no pathological or morphological alteration.

Exclusion Criteria:

* untreated periodontitis;
* previous surgery on the palate;
* history of poor wound healing;
* systemic diseases and/or coagulations disorders;
* pregnant or lactating;
* smoking or marijuana use (non-smoker status verified by exhaled air carbon monoxide as previously described);
* medications affecting periodontal status (e.g. phenytoin, calcium channel blockers and cyclosporine);
* therapy with anticoagulants, nonsteroidal anti-inflammatory drugs, corticosteroids, or any drug interfering with the healing process during the previous six months;
* contraindication to receiving any of the active components of the antimicrobial gel.

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Estimated)
Dates: Start 2024-12-22 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Color Match (CM) | CM will be evaluated on post-operative days 1, 3, 7, 14, 21 and 30
  CM will be evaluated comparing color of the adjacent and opposite sides again using VAS scores from 0 (no CM) to 10 (excellent CM)

SECONDARY OUTCOMES:
Healing Index (HI) | HI will be assessed on post-operative days 1, 3, 7, 14, 21 and 30
  The Pippi modification of the Landry index will be calculated as the sum of seven parameters, each of them will be observed clinically and then will receive a dichotomic score (0/1): a total score of 7 will be associated with better healing process. The assessed parameters will be the following:
  * Presence or absence of redness;
  * Presence or absence of granulation tissue;
  * Presence or absence of suppuration;
  * Presence or absence of swelling;
  * Degree of tissue re-epithelization (partial or complete);
  * Presence or absence of bleeding;
  * Presence or absence of pain on palpation.
Secondary Healing Classification (SHC) | SHC will be assessed on post-operative days 1, 3, 7, 14, 21 and 30
  This Classification is composed by 3 classes (I,II,III) and 3 sub-classes (a,b,c). Class I and Sub-class a are associated with complete wound closure and optimal healing.
Complete epithelization (CE) | CE will be assessed on post-operative days 1, 3, 7, 14, 21 and 30.
  CE will be assessed clinically after direct visualization via inspection supported by means of clinical photographs taken at each post-surgical visit to provide insight into the differences among patients across all groups. CE will recorded as dichotomous scoring by a clinical investigator masked to all groups as "yes" or "no" according to inspectional evaluation of surface characteristics and reflection as well as clarity and distinctness of wound outline. If the epithelial barrier is intact and if distinction of a demarcation line is unclear when assessing the edges, CE was scored as "yes."
Oral Health Impact Profile-14 (OHIP-14) | It will be evaluated at baseline and on post-operative days 1, 3, 7, 14, 21 and 30
  Participants will be also asked to complete the OHIP-14 questionnaire.
Functional Pain Scale (FPS) | It will be assessed on post-operative days 1, 3, 7, 14, 21 and 30.
  To assess pain experience and questions related to number of analgesics (NA) consumed and postoperative complications experienced during the first 14 days.
Swelling | It will be assessed on post-operative days 1, 3, 7, 14, 21 and 30.
  It will be also evaluated using VAS . VAS: from 0 (no swelling) to 10 (maximal swelling)
Burning sensation | It will be assessed on post-operative days 1, 3, 7, 14, 21 and 30.
  It will be also evaluated using VAS . VAS: from 0 (no burning sensation) to 10 (maximal burning sensation)
Discomfort | It will be assessed on post-operative days 1, 3, 7, 14, 21 and 30.
  It will be also evaluated using VAS . VAS: from 0 (no discomfort) to 10 (maximal discomfort)

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza University of Rome, Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: No